CLINICAL TRIAL: NCT05717790
Title: Nimotuzumab Combined With Induction Chemotherapy Plus Chemoradiation and Adjuvant Therapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Concurrent and Adjuvant Nimotuzumab Combined With Induction Chemotherapy Plus Chemoradiation in Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fourth Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: People's Hospital of Baise (Unknown); Second Affiliated Hospital of Guangzhou Medical University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Guilin Medical University, China (Other); LiuZhou People's Hospital (Other); The First People's Hospital of Qinzhou (Unknown); Wuzhou Red Cross Hospital (Other); Youjiang Medical College for Nationalities (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZLK3815405
Record Dates: First submitted 2022-12-24; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V8 Stage
Keywords: Nimotuzumab; Nasopharyngeal Carcinoma; Induction Chemotherapy; Chemoradiation; Adjuvant Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab; Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Nimotuzumab arm (Experimental): Patients will receive induction chemotherapy with nimotuzumab (200mg/w,weekly plus gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 2 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) will be given. Concurrent nimotuzumab (200mg/w,weekly, 6-7 weeks) and cisplatin (100mg/m2,every 3 weeks for 3cycles )will be administered during IMRT. After 4-6 weeks of the completion of IMRT, adjuvant nimotuzumab (200mg ) will be given every 3 weeks for 8 cycles.
  Interventions: Drug: Nimotuzumab; Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy
- Control (Active Comparator): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 2 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) will be given. Concurrent nimotuzumab (200mg/w,weekly, 6-7 weeks) and cisplatin (100mg/m2,every 3 weeks for 3cycles )will be administered during IMRT.
  Interventions: Drug: Nimotuzumab; Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — Drug: Nimotuzumab Experimental: Nimotuzumab arm Induction chemotherapy:Nimotuzumab 200mg will be given weekly for 6 cycles, started on day 1 of induction chemotherapy.
  Concurrent chemotherapy: Nimotuzumab 200mg/week in concurrent with IMRT. Adjuvant therapy: Nimotuzumab (200mg ) will be given every 3 weeks for 8 cycles.
  Active Comparator: Control Nimotuzumab 200mg/week in concurrent with IMRT .
  Other Names: h-R3; BIOMAb EGFR
Drug: Gemcitabine — Gemcitabine as induction chemotherapy, 1000 mg/m2 day 1, 8 per cycle, every 3 weeks for 2 cycles
  Other Names: GEM
Drug: Cisplatin — Cisplatin as induction chemotherapy, 80 mg/m2 day 1 per cycle, every 3 weeks for 2 cycles.
  Cisplatin as concurrent chemotherapy, 100 mg/m2 day 1 per cycle, every 3 weeks for 3 cycles.
  Other Names: DDP
Radiation: Intensity-modulated radiotherapy — Definitive IMRT of 68-78 Gy, 30-33 fractions, 5 fractions/week, 1 fraction/day
  Other Names: IMRT

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Nimotuzumab has been granted approval for use in squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal cancer in different countries. This is a multi-center, randomized controlled trial, with the purpose to evaluate the therapeutic efficacy and safety of nimotuzumab combined with induction chemotherapy plus chemoradiation and adjuvant therapy in locoregionally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 70.
2. Pathological type: non-keratinizing carcinoma (World Health Organization criteria).
3. Diagnosed with LANPC (stage III-IV, except for patients with T3N0)) according to the 8th edition clinical staging system of the American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC].
4. ECOG performance score: 0 to 1.
5. Primary lesions can measurable.
6. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
7. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and creatinine clearance rate ≥ 50 ml/min (Cockcroft-Gault formula).
8. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Primary lesions or lymph node have been operated (except of operation for biopsy).
2. Previous Received other anti EGFR monoclonal antibody treatment;Previous chemotherapy or immunization therapy.
3. Other malignant tumor.
4. Participation in other interventional clinical trials within 1 month.
5. History of Serious lung or heart disease.
6. Pregnant or breast-feeding women and women who refused to take contraceptive method.
7. Drug abuse or alcohol addiction.
8. History of serious allergic or allergy.
9. Refused or can't signed informed consent form.
10. Other patients who are considered ineligible for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
overall survival(OS) | 5 years
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive.OS will be measured by the Method of Kaplan and Meier.

SECONDARY OUTCOMES:
Tumor control probability (TCP) | 5 years
  Tumor control probability is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: at least 30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Disease-free survival(DFS) | 5 years
  DFS is defined as the time from randomization to the first documented disease progression or death due to disease progression per RECIST 1.1. DFS will be measured by the Method of Kaplan and Meier.
Locoregional failure-free survival(LRRFS) | 5 years
  LRRFS is defined as the time from randomization to the date of locoregional relapse per RECIST 1.1. LRRFS will be measured by the Method of Kaplan and Meier.
Distant Metastasis-free survival(DMFS) | 5 years
  DMFS is defined as the time from randomization to the date of first distant metastasis. DMFS will be measured by the Method of Kaplan and Meier.
Incidence rate of investigator-reported adverse events (AEs) | 5 years
  Analysis of investigator-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0 and radiation therapy oncology group (RTOG) toxicity criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 5 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, MD, Principal Investigator — The Fourth Affiliated Hospital of Guangxi Medical University
Locations (9):
- China (9):
  - People's Hospital of Baise, Baise City, Guangxi
  - Affiliated Hospital of Youjiang Medical University for Nationalities, Baise City, Guangxi
  - Guilin Medical University, China, Guilin, Guangxi
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi
  - the Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi
  - Second Affiliated Hospital of Guangzhou Medical University, Nanjing, Guangxi
  - The First People's Hospital of Qinzhou, Qinzhou, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - Liuzhou People's Hospital, Liuchow, Other (Non U.s.)

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: For 2 years started from 12 months after publication of the primary trial report.
Access Criteria: Authoritative researchers who provide a methodologically sound proposal for individual participant data meta-analysis.